CLINICAL TRIAL: NCT06098014
Title: Safety & Efficacy of Thalidomide in Children With Transfusion Dependent Thalassemia: a Quasi Randomized Control Trial in a Tertiary Care Hospital in Bangladesh
Brief Title: Safety & Efficacy of Thalidomide in Children With Transfusion Dependent Thalassemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Md. Mehedi Hasan, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4280
Record Dates: First submitted 2023-10-12; First posted 2023-10-24 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Transfusion-dependent Thalassemia
Keywords: Thalidomide,; Thalassemia; Children
MeSH Terms: conditions — Thalassemia | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thalidomide group (Active Comparator): Thalidomide group
  Interventions: Drug: Thalidomide Capsules
- Placebo group (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide Capsules — To see safety and efficacy of Thalidomide in Transfusion depended thalassemia
  Arms: Thalidomide group
Drug: Placebo — compare with Thalidomide
  Arms: Placebo group

SUMMARY:
Transfusion Dependent Thalassemia (TDT) is emerging as a global public health concern. Hemopoietic stem cell transplantation (HSCT) is the only curative treatment. But its adoption is limited due to lack of Human leukocyte antigen (HLA) matched donor, experienced centers and high initial cost. So, researches are going on in search of an effective, safe, easily available treatment option. Thalidomide a Fetal Hemoglobin (HbF) inducing drug shown to be effective in treatment of TDT patients in few case reports and small scale prospective and retrospective studies. However, most of these researches were done in adolescent and adult population. No randomized control trial was done to determine the safety and efficacy of Thalidomide in TDT children. So, this study will predict the safety and efficacy of Thalidomide in TDT children and will play an important role in planning a cost effective and affordable treatment option for TDT children.

This single centered non blinded quasi randomized clinical trial will be conducted at the Department of Pediatric Hematology and Oncology in Bangabandhu Sheikh Mujib Medical University (BSMMU), Bangladesh for one year of period. The objective of this study is to assess the safety and efficacy of Thalidomide in TDT children 30 transfusion dependent thalassemia children of 3-18 years old will be included.

This study will involve minimum physical risk to the patient. Written informed consent will be taken from parents or study subjects after brief explanation of the purpose and procedure. They will also be informed about the freedom to participate or not to participate at any time. Privacy and confidentiality will be safe guarded. History regarding age, sex, height, weight of these patients will be taken. Through physical examinations and laboratory investigations including complete blood count (CBC), Hb electrophoresis, serum Ferritin, serum creatinine, serum glutamic pyruvic transaminase (SGPT), serum lactate dehydrogenase (LDH) will be done.

Data will be collected in a predesigned questionnaire and will be kept confidential. Statistical analysis will be done using the statistical package for social science (SPSS) software .

DETAILED DESCRIPTION:
Study design: Quasi-randomized controlled tria

Period of Study: From March 2023 to February 2023

Place of study:

Department of Pediatric Hematology & Oncology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Bangladesh.

Study Population:

TDT patients of either gender and 3-18 years of age attending in the Department of Pediatric Hematology and Oncology, Bangabandhu Sheikh Mujib Medical University, Dhaka and will receive Thalidomide during the study period.

Sample size will be calculated by using following formula:

((u+v)^2 (σ₁²+σ₀²))/((μ₁-μ₀)²) Here, u = .842 (if power= 80%) v = 1.96 (if significance level= 5%) μ₀ (mean Hb level before treatment with Thalidomide) = 71 μ₁ (mean Hb level in after treatment with Thalidomide) = 95 σ₀ = assumed population standard deviation for Placebo group = 30 σ₁ = assumed population standard deviation for Thalidomide group = 30

Calculated sample size is:

((u+v)^2 (σ₁²+σ₀²))/((μ₁-μ₀)²)

* (1.96+0.842)2 ( 30² +30²)/ (24)2

= 24.5 ~25

Group sample sizes of 25 in each group, considering 10% drop out it may increase up to 30 as some cases may be lost to follow up during study period.

So, sample size will be 30+30 = 60.

Sampling technique:

From the date of start of study, patient will be selected purposively by inclusion and exclusion criteria during the desired study period. The patients will be randomized 1:1 to receive placebo or thalidomide. Block or restricted randomization will be used to select the intervention group and control. All odd number patients (1,3,7…) will be considered as block & will be assigned to intervention group by lottery and then all even number patients (2,4,6…) will be assigned to the other group.

Data collection procedure:

This study will be conducted in the Department of Pediatric Hematology and Oncology, Bangabandhu Sheikh Mujib Medical University (BSMMU). Children aged 3 to 18 years of both sexes diagnosed as TDT visiting the hematology out patient department (OPD) between March 2023 to February 2024 will be included in this study. Informed written consent from the patients or parents or guardians will be obtained at the time of study enrollment.

After recruitment, subjects will be randomly divided into two groups according to the Thalidomide therapy as follows:

1. Experimental Group: Patients who will receive Thalidomide along with regular drugs.
2. Control Group: Patients who will receive placebo with other regular drugs are considered as in the control group.

Data will be collected using a preformed data collection sheet (questionnaire). Demographic data such as age, sex, socio-economic status, family history of thalassemia will be collected from guardian or parents. Medical data regarding age, sex, age at first transfusion, red cell transfusion in last 1 year will be compiled. Clinical information such as pallor, pulse, blood pressure, respiratory rate, spleen size and other systemic clinical parameters will be taken.

Thalidomide and placebo will be given to randomly selected patients as per inclusion criteria attending in the outpatient department. The instruction will be given by the principal investigator according to study design.

Patients diagnosed with transfusion-dependent thalassemia will be randomized to receive placebo or Thalidomide treatment at a dose of 2-5 mg/kg/day.

The initial evaluation will be performed before the patients started Thalidomide. Patients will get transfusion with red blood cells at 10 ml/kg at any time during the study period if their Hb level < 70 g/L. The patients are followed up every 14 days for the first 12 weeks, and every 3 months thereafter. The efficacy will be evaluated after 12 weeks of treatment. Additionally, in patients with an obvious elevation in Hb who are free from blood transfusions for at least 6 weeks, the original treatment will be continuously administered for further evaluation. When the last patient is enrolled and completes their first 12 weeks of follow-up, the placebo-controlled period of the study will end.

Each evaluation will be included in a data collection sheet that will record crucial information such as the evaluation number, age, sex, type of diagnosis, Hb level, transfusion requirement etc. All participants will be asked to report any adverse reactions and will be questioned about adverse events during study visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as transfusion dependent thalassemia
* Age ranged from 3-18 years
* Blood transfusion for more than 1 year.

Exclusion Criteria:

* Active systemic illness,
* Abnormal liver and kidney functions;
* Severe cardiopulmonary or cerebrovascular diseases;
* Recent fracture or recent major surgery
* Use of drugs that might affect Hb levels 3 months before enrollment;
* Any bleeding disorder .

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
change in Hb level | 12 weeks after treatment initiation.
  gm/dl

SECONDARY OUTCOMES:
blood transfusion frequency | 3 months from initiation of treatment
  time
change in Hb F | 3 months after initiation of treatment
Change in s. Ferritin level | 3 months after initiation of treatment
  ng/mL
Adverse effect | 3 months after initiation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2025

REFERENCES:
- [Background] Fard AD, Hosseini SA, Shahjahani M, Salari F, Jaseb K. Evaluation of Novel Fetal Hemoglobin Inducer Drugs in Treatment of beta-Hemoglobinopathy Disorders. Int J Hematol Oncol Stem Cell Res. 2013;7(3):47-54. PMID 24505535
- [Background] Farmakis D, Porter J, Taher A, Domenica Cappellini M, Angastiniotis M, Eleftheriou A. 2021 Thalassaemia International Federation Guidelines for the Management of Transfusion-dependent Thalassemia. Hemasphere. 2022 Jul 29;6(8):e732. doi: 10.1097/HS9.0000000000000732. eCollection 2022 Aug. PMID 35928543
- [Background] Fozza C, Pardini S, Giannico DB, Targhetta C, Di Tucci AA, Dessalvi P, Angelucci E, Dore F. Dramatic erythroid response to low-dose thalidomide in two patients with transfusion independent thalassemia and severe post-transfusional alloimmune hemolysis. Am J Hematol. 2015 Jul;90(7):E141. doi: 10.1002/ajh.24030. No abstract available. PMID 25850682
- [Background] Hossain MS, Raheem E, Sultana TA, Ferdous S, Nahar N, Islam S, Arifuzzaman M, Razzaque MA, Alam R, Aziz S, Khatun H, Rahim A, Morshed M. Thalassemias in South Asia: clinical lessons learnt from Bangladesh. Orphanet J Rare Dis. 2017 May 18;12(1):93. doi: 10.1186/s13023-017-0643-z. PMID 28521805
- [Background] Jain M, Chakrabarti P, Dolai TK, Ghosh P, Mandal PK, Baul SN, De R. Comparison of efficacy and safety of thalidomide vs hydroxyurea in patients with Hb E-beta thalassemia - a pilot study from a tertiary care Centre of India. Blood Cells Mol Dis. 2021 May;88:102544. doi: 10.1016/j.bcmd.2021.102544. Epub 2021 Feb 3. PMID 33610115
- [Background] Lu Y, Wei Z, Yang G, Lai Y, Liu R. Investigating the Efficacy and Safety of Thalidomide for Treating Patients With ss-Thalassemia: A Meta-Analysis. Front Pharmacol. 2022 Jan 11;12:814302. doi: 10.3389/fphar.2021.814302. eCollection 2021. PMID 35087410
- [Background] Masera N, Tavecchia L, Capra M, Cazzaniga G, Vimercati C, Pozzi L, Biondi A, Masera G. Optimal response to thalidomide in a patient with thalassaemia major resistant to conventional therapy. Blood Transfus. 2010 Jan;8(1):63-5. doi: 10.2450/2009.0102-09. No abstract available. PMID 20104280
- [Background] Rachmilewitz EA, Giardina PJ. How I treat thalassemia. Blood. 2011 Sep 29;118(13):3479-88. doi: 10.1182/blood-2010-08-300335. Epub 2011 Aug 2. PMID 21813448
- [Background] Shah FT, Sayani F, Trompeter S, Drasar E, Piga A. Challenges of blood transfusions in beta-thalassemia. Blood Rev. 2019 Sep;37:100588. doi: 10.1016/j.blre.2019.100588. Epub 2019 Jul 6. PMID 31324412
- [Background] Taher A, Vichinsky E, Musallam K, Cappellini MD, Viprakasit V, authors. Weatherall D, editor. Guidelines for the Management of Non Transfusion Dependent Thalassaemia (NTDT) [Internet]. Nicosia (Cyprus): Thalassaemia International Federation; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK190453/ PMID 24672826
- [Background] Thompson AA, Walters MC, Kwiatkowski J, Rasko JEJ, Ribeil JA, Hongeng S, Magrin E, Schiller GJ, Payen E, Semeraro M, Moshous D, Lefrere F, Puy H, Bourget P, Magnani A, Caccavelli L, Diana JS, Suarez F, Monpoux F, Brousse V, Poirot C, Brouzes C, Meritet JF, Pondarre C, Beuzard Y, Chretien S, Lefebvre T, Teachey DT, Anurathapan U, Ho PJ, von Kalle C, Kletzel M, Vichinsky E, Soni S, Veres G, Negre O, Ross RW, Davidson D, Petrusich A, Sandler L, Asmal M, Hermine O, De Montalembert M, Hacein-Bey-Abina S, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in Patients with Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2018 Apr 19;378(16):1479-1493. doi: 10.1056/NEJMoa1705342. PMID 29669226
- [Background] Weatherall DJ. The Evolving Spectrum of the Epidemiology of Thalassemia. Hematol Oncol Clin North Am. 2018 Apr;32(2):165-175. doi: 10.1016/j.hoc.2017.11.008. PMID 29458724
- [Background] Wolman IJ, Ortolani M. Some clinical features of Cooley's anemia patients as related to transfusion schedules. Ann N Y Acad Sci. 1969 Nov 20;165(1):407-14. doi: 10.1111/j.1749-6632.1969.tb27811.x. No abstract available. PMID 5260163
- [Background] Yassin AK. Promising Response to Thalidomide in Symptomatic beta-Thalassemia. Indian J Hematol Blood Transfus. 2020 Apr;36(2):337-341. doi: 10.1007/s12288-019-01231-5. Epub 2019 Nov 18. PMID 32425386
- [Result] Aerbajinai W, Zhu J, Gao Z, Chin K, Rodgers GP. Thalidomide induces gamma-globin gene expression through increased reactive oxygen species-mediated p38 MAPK signaling and histone H4 acetylation in adult erythropoiesis. Blood. 2007 Oct 15;110(8):2864-71. doi: 10.1182/blood-2007-01-065201. Epub 2007 Jul 9. PMID 17620452
- [Result] Aguilar-Lopez LB, Delgado-Lamas JL, Rubio-Jurado B, Perea FJ, Ibarra B. Thalidomide therapy in a patient with thalassemia major. Blood Cells Mol Dis. 2008 Jul-Aug;41(1):136-7. doi: 10.1016/j.bcmd.2008.03.001. Epub 2008 Apr 24. No abstract available. PMID 18439858
- [Result] Bou-Fakhredin R, De Franceschi L, Motta I, Cappellini MD, Taher AT. Pharmacological Induction of Fetal Hemoglobin in beta-Thalassemia and Sickle Cell Disease: An Updated Perspective. Pharmaceuticals (Basel). 2022 Jun 16;15(6):753. doi: 10.3390/ph15060753. PMID 35745672
- [Result] Cappellini MD, Porter JB, Viprakasit V, Taher AT. A paradigm shift on beta-thalassaemia treatment: How will we manage this old disease with new therapies? Blood Rev. 2018 Jul;32(4):300-311. doi: 10.1016/j.blre.2018.02.001. Epub 2018 Feb 12. PMID 29455932
- [Result] Chen JM, Zhu WJ, Liu J, Wang GZ, Chen XQ, Tan Y, Xu WW, Qu LW, Li JY, Yang HJ, Huang L, Cai N, Wang WD, Huang K, Xu JQ, Li GH, He S, Luo TY, Huang Y, Liu SH, Wu WQ, Lu QY, Zhou MG, Chen SY, Li RL, Hu ML, Huang Y, Wei JH, Li JM, Chen SJ, Zhou GB. Safety and efficacy of thalidomide in patients with transfusion-dependent beta-thalassemia: a randomized clinical trial. Signal Transduct Target Ther. 2021 Nov 18;6(1):405. doi: 10.1038/s41392-021-00811-0. PMID 34795208
- [Result] Costa E, Cappellini MD, Rivella S, Chilin A, Alessi E, Riccaboni M, Leufkens HGM, Luzzatto L. Emergent treatments for beta-thalassemia and orphan drug legislations. Drug Discov Today. 2022 Nov;27(11):103342. doi: 10.1016/j.drudis.2022.103342. Epub 2022 Sep 1. PMID 36058507